CLINICAL TRIAL: NCT03814928
Title: Recovery After Hip Fracture: A Novel Online Intervention for Caregivers
Brief Title: Caregivers' eCourse for Recovery After Hip Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H18-01409
Record Dates: First submitted 2018-05-21; First posted 2019-01-24 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Hip Fractures; Family
Keywords: education; caregivers; eCourse; feasibility
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: feasibility study with the general public, older adults, health providers, and family caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregivers eCourse (Experimental): Education post-hip fracture delivered via eCourse.
  Interventions: Behavioral: Caregivers eCourse

INTERVENTIONS:
Behavioral: Caregivers eCourse — Investigators will request that family/caregivers/general public watch a self-paced (60-90 minutes) online e-learning training session for recovery after hip fracture.

SUMMARY:
In this two part study, we will seek 1. general feedback on the feasibility of an online education and skill development program for family/caregivers of older adults recovering from a surgically repaired low-trauma hip fracture. We will also 2. test its feasibility and acceptability with family caregivers.

DETAILED DESCRIPTION:
This is a cross-sectional mixed methods study to obtain feedback from health providers and family caregivers on eCourse for the post-hip fracture period. For participants who access the course via the PI's website, participants will only be asked to provide feedback on the content, layout, and delivery of the eCourse.

ELIGIBILITY:
Inclusion Criteria:

* Family/caregivers of older adults with hip fracture, health providers, older adults, and/or general public

Exclusion Criteria:

* Adults less than 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
eCourse Acceptibility | Day 1
  Participants will be asked to rate (using a Likert scale 1 to 10) perceptions of acceptability of the (1) delivery mode and (2) program. All three questions are rate from 1 (lowest) - 10 (highest). A higher score is better.
eCourse Feasibility | Day 1
  Participants will be asked to rate (using a Likert scale 1 to 10) perceptions of feasibility of the (1) delivery mode and (2) program. All three questions are rate from 1 (lowest) - 10 (highest). A higher score is better.
eCourse Satisfaction | Day 1
  We will ask people to rate their satisfaction with the eCourse [1 (not satisfied) to 10 (very satisfied)]. The higher the score the better.
eCourse Usefulness | Day 1
  We will ask people to rate their perception of the usefulness for the eCourse [1 (not useful) to 10 (very useful)]. The higher the score the better.
Modified Computer Self-Efficacy Scale | Day 1
  Questionnaires will assess participants' perceptions of self-efficacy (Modified Computer Self-Efficacy Scale) for using a computer and the online program. Scale of 1-10, 1 (not at all confident) - 10 (completely confident). The higher the score the better.
Unified Theory of Acceptance and Use of Technology 2 | Day 1
  Questionnaires will assess participants' perceptions on technology usability (Unified Theory of Acceptance and Use of Technology 2). Participants will rate on a scale of 1-5, how much they disagree/agree with statements. 1 (strongly disagree) - 5 (strongly agree)
Caregivers' eCourse semi-structured interviews | Day 1
  We will conduct semi-structured interviews with caregivers to further explore perceptions and experience with eCourse and caregiving after hip fracture.
Feedback on eCourse for participants who enrol via the PI's website: PEMAT | Day 1
  Patient Education Materials Assessment Tool (PEMAT) to evaluate the understandability and actionability of the material in our eCourse.

SECONDARY OUTCOMES:
Caregiver Strain Index | Day 1
  Ten questions on factors affected by caregiving with a yes or no response.
EQ5D-5L (health-related quality of life) | Day 1
  Five domains of questions with five responses each. Calculate an index of 0 (lowest) - 1 (highest). There is also a Visual Analogue Scale [1 (worse health) - 100 (best health)]
ICECAP-O (general quality of life) | Day 1
  Five domains of questions with four responses each. Calculate an index of 0 (lowest) - 1 (highest).

CONTACTS AND LOCATIONS:
Locations (1):
- UBC, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No